CLINICAL TRIAL: NCT03581929
Title: Randomized Controlled Trial to Evaluate the Efficacy of a Food Supplement, in Subjects With Mild Cognitive Impairment (MCI)
Brief Title: Efficacy of MEMORMAX in Subjects With MCI
Acronym: ABO-MEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: Latis S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: MEMORMAX
Record Dates: First submitted 2018-05-15; First posted 2018-07-10 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Dementia; Memormax; Food Supplement; Microbiota
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind from Day 0 to Day 180. Open Label from Day 181 to Day 360.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memormax (Experimental): 2 vials / day of Memormax from Day 0 to Day 180. At the end of the blinded phase (Day 0-180), all patients will receive 2 vials / day of Memormax from Day 181 to Day 360.
  Interventions: Dietary Supplement: Memormax
- Placebo (Placebo Comparator): 2 vials / day of Placebo from Day 0 to Day 180. At the end of the blinded phase (Day 0-180), all patients will receive 2 vials / day of Memormax from Day 181 to Day 360.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Memormax — Memormax is a food supplement indicated to support cognitive functions thanks to the Melissa officinalis; it also contains lyophilized Royal Jelly, Blueberry extract and Blueberry juice.
  Arms: Memormax
Other: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blinded placebo for the first 6 months of treatment in subjects with mild cognitive impairment. Open-label treatment, with all subjects receiving active treatment, for the next 6 months of study.

DETAILED DESCRIPTION:
Patients are enrolled in the department of Geriatria, Azienda Ospedaliera di Perugia. The group of this pilot project will include 50 subjects. All the volunteers who, in compliance with the inclusion and exclusion criteria, will be available for follow-up at twelve months and are able to give informed written consent guaranteeing adherence to the treatment will be enrolled in the study.

The study involves the collection of clinical data acquired as part of routine assessments for the type of subject included in this research project.

Visit 1 baseline: day 1 (time 0) Upon enrollment, all subjects, for whom informed consent will be obtained, will undergo a medical examination for an overall assessment of the state of health. In all subjects, a careful family, pathological and pharmacological anamnesis will be collected, data on the habits of life (nutrition, smoking, exercise) will be collected through a specific questionnaire and the main anthropometric parameters will be evaluated (weight, height,body mass index, waist / hip ratio) and the risk of development of cognitive impairment through the Brief Late-life Dementia Risk Index (Barnes et al., 2014).

The clinical examination will be completed by a standard assessment for the hematobiochemical and urinalysis examinations.

The results of the tests and of the tests carried out for the diagnosis of MCI, according to the clinical practice of the center, will be collected and used as baseline values, up to one month before entry into the study.

In addition, some physical performance tests will be performed (hand grip evaluation, timed up and go, SPPB, frailty index, bioimedenzometry (BIA)). The results of the following tests and examinations carried out for the diagnosis of MCI will be collected, in the month before entry into the study: ECG, physical performance test (through evaluation of ADL, IADL), cognitive performance test (FCSRT, MMSE, ACE -R, Digit Span forward, Digit Span back, Trail Making A and B, Babcock story, Rey test, Raven test, Token test, verbal fluency test, prose memory, copy of drawings, verbal reviews), tests for the presence of behavioral disorders (Neuropsychiatric Inventory scale, NPI) and mood (Geriatric Depression Scale, GDS), Cognitive Reserve Index (CRI) (Nucci et al., 2012) in order to verify if the cognitive reserve could somehow to explain the variability found.

At this visit the patient will be randomized to receive one of the following products daily for 6 months:

A) Memormax, 2 vials / day B) Placebo, 2 vials / day. Each patient will receive a supply of 30 packs of 12 vials each of Memormax or Placebo. Finally, the material for stool collection will be delivered to the patients. Patients will then be instructed to not start treatment in the study before collecting the faecal sample. This sample must be returned to the center in the days immediately following the visit 1.

Visit 2 - time 6 months (± 5 days) After 6 months all subjects will be subjected to medical evaluation (functional and cognitive), venous blood sampling, urine test and ECG control. Any changes in concomitant therapies and any adverse events will be recorded. Unused and used vials will be collected for accounting and verification of treatment compliance. All the subjects in the study (n = 50) will receive for the next 6 months only Memormax, according to an open study design. Each patient will receive a supply of 30 packs of 12 vials each of Memormax.

Visit 3 - time 12 months (end of study / premature termination of the study) At twelve months, all subjects will be subjected to medical evaluation (functional and cognitive), peripheral venous blood sampling, urine test and ECG control. Any changes in concomitant therapies and any adverse events will be recorded. Unused and used vials will be collected for accounting and verification of treatment compliance. In the event of premature termination of the study by a patient, at any time after the start of treatment, all assessments scheduled for Visit 3 should be made, considering the visit itself as the conclusion of the study for that patient. It is specified that in the follow-up evaluations (6 and 12 months) the parallel versions of the instruments used at the baseline will be used to avoid learning effects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mild cognitive impairment, according to operational criteria for defining Mild Cognitive Impairment (MCI) (Albert et al, 2011): change in cognitive status, mild deficit in one or more cognitive domains, normal ability to perform activities in daily life or slight deficits not related to cognitive reasons, absence of dementia;
* MMSE≥24
* Good level of functional autonomy: ADL ≥ 5 / 6, IADL ≥ 4 / 8 for male subjects, ≥ 6/8 for female subjects, SPPB with score ≥ 9; Walk speed test in 6 meters ≥ 1 m / s;
* Written informed consent of the patient.

Exclusion Criteria:

* Subjects with malignant neoplasia in progress or diagnosed within 5 years;
* Subjects with active infections or autoimmune pathogenesis diseases (eg sclerosis, Chron, polymyalgia);
* Subjects diagnosed with neurodegenerative disease in pharmacological treatment (eg Parkinson's disease)
* Subjects with psychiatric conditions (eg psychosis, depression, schizophrenia)
* Subjects in pharmacological treatment for urinary incontinence
* Subjects with involuntary weight loss> 5 kg in the last twelve months;
* Subjects with chronic renal failure ≥ stage III K-DOQI;
* Subjects with clinically significant liver disease (AST / SGOT, ALT / SGPT> 2 upper limits)
* Subjects with severe hearing, vision, speech or walking disabilities;
* Geriatric Depression Scale (Geriatric Depression Scale)> 4 out of 15 items;
* Consumption in the two months prior to the baseline assessment of supplements containing omega-3 fatty acids or foods containing fish oil, foods for special medical purposes (AFMS);
* Use in the month prior to baseline assessment of: atropine, scopolamine, tolterodine, iosciamin, biperidene, benzotropin, oxybutynin, antipsychotics, vitamins B, C and / or> at 200% of the suggested daily dose, highly energetic nutritional supplements and / or proteins, other products under experimentation;
* Alcohol abuse.
* Use of antibiotics in the two months preceding the baseline assessment;
* Regular use of probiotics, fiber supplements or laxative

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Memormax efficacy on global cognitive performance (FCRST). | Day 0-180
  Effect of Memormax on global cognitive performance in patients with mild Mild Cognitive Impairment (MCI) after a 6 months treatment and compared to placebo (T0-T6), measured by the FREE AND CUED SELECTIVE REMINDING TEST (FCRST)
Memormax efficacy on global cognitive performance (ACE-R). | Day 0-180
  Effect of Memormax on global cognitive performance in patients with mild Mild Cognitive Impairment (MCI) after a 6 months treatment and compared to placebo (T0-T6), measured by the ADDENBROOKE'S COGNITIVE EXAMINATION (ACE-R) tests.
Effect of Memormax on global cognitive performance across the entire population (FCRST) | Day 181-360
  To evaluate the effect of Memormax on global cognitive performance across the entire population studied in a 6-month open-label extension phase (T6-T12), measured by the FCSRT
Effect of Memormax on global cognitive performance across the entire population (ACE-R) | Day 181-360
  To evaluate the effect of Memormax on global cognitive performance across the entire population studied in a 6-month open-label extension phase (T6-T12), measured by the ACE-R

SECONDARY OUTCOMES:
variations of the main parameters of cognitive performance (MMSE) | Day 0-180-360
  Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. The MMSE test includes simple questions that are valuated using point subscales that are summed to have a maximunm of 30 points; the administration of the test takes between 5 and 10 minutes and cognitive functions of each patient are examinated as reported below; Orientation to time (0-5 points), Orientation to place (0-5 points), Registration (0-3 points), Attention and calculation (0-5 points), Recall (0-3 points), Language and Praxis (0-9 points).
  If the score is greater than or equal to 24, patient has a normal cognition. Below 24 points, we can indicate a severe cognitive impairment (≤9 points), a moderate cognitive impairment (10-18 points) and a mild cognitive impairment (19-23 points). For these reasons, higher values represent a better outcome
variations of the main parameters of cognitive performance (Digit Span) | Day 0-180-360
  A digit-span task is used to measure working memory's number storage capacity. Participants see or hear a sequence of numerical digits and are tasked to recall the sequence correctly, with increasingly longer sequences being tested in each trial. The participant's span is the longest number of sequential digits that can accurately be remembered.measured with further tests that explore multiple cognitive functions compared to evaluations as primary objectives.
variations of the main parameters of cognitive performance (Trail Making) | Day 0-180-360
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
variations of the main parameters of cognitive performance (Babcock) | Day 0-180-360
  Babcock Story Recall Test (BSRT; Babcock &. Levy, 1940) is a verbal memory measure in which participants are read a brief story and asked to provide a summary of the story.
variations of the main parameters of cognitive performance (Rey Test) | Day 0-180-360
  The Rey 15-Item test is a test designed by Rey (1964) to detect malingering.
variations of the main parameters of cognitive performance (Raven Test) | Day 0-180-360
  Raven's Progressive Matrices (often referred to simply as Raven's Matrices) or RPM is a nonverbal group test typically used in educational settings. It is usually a 60-item test used in measuring abstract reasoning and regarded as a non-verbal estimate of fluid intelligence
variations of the main parameters of cognitive performance (Token Test) | Day 0-180-360
  The original TT tested auditory verbal memory by having the subject point to tokens of 5 different colors, 2 shapes (circle, squares), and 2 sizes (small, large), in response to commands such as "touch the blue circle" (a one dimensional command, or 1-D, since the tokens differ only by color), or "touch the yellow square and the red circle" (a two dimensional command, or 2-D, since the tokens differ by color and/or shape), or "touch the small red circle and the large green square" (a three dimensional command, or 3-D, since the tokens differ by size, and/or color and/or shape).
variations of the main parameters of cognitive performance (Verbal Fluency) | Day 0-180-360
  Verbal fluency tests are a kind of psychological test in which participants have to produce as many words as possible from a category in a given time (usually 60 seconds)
variations of the main parameters of cognitive performance (NEPSY-II) | Day 0-180-360
  NEPSY-II is the only single measure that allows the clinician to create a tailored assessment across the following domains: Executive functioning, Attention Language, Memory and learning, Sensorimotor functioning, Social perception, Visuospatial processing. The results provide information relating to typical childhood disorders, which can lead to accurate diagnosis and intervention planning for success in school and at home
variations of the main parameters of cognitive performance (NPI) | Day 0-180-360
  Standard Neuropsychiatric Inventory-Questionnaire providing a brief assessment of neuropsychiatric symptomatology in routine clinical practice settings.
  Standard Neuropsychiatric Inventory-Questionnaire, analyzes the Severity of the symptoms present within the last month on a 3-point scale: 1 (mild), 2 (moderate), 3 (severe). This questionnaire analyzes also the distress on a 5-points scale described below:
  0 = Not distressing at all
  1. = Minimal
  2. = Mild
  3. = Moderate
  4. = Severe
  5. = Extreme or Very Severe
variations of the main parameters of cognitive performance (GDS) | Day 0-180-360
  The Geriatric Depression Scale (GDS) is a 30-item self-report assessment used to identify depression in the elderly. Patients have to answer, with YES (0 point) or NO (1 point), to the questions and the following general cutoff may be used to qualify the severity:
  normal 0-9, mild depressives 10-19, severe depressives 20-30.
variations of the main parameters of cognitive performance (Cognitive Reserve Index) | Day 0-180-360
  The cognitive Reserve Questionnaire (CRIq) is an instrument for measuring the cognitive reserve of an individual by means of the compilation of information relating to his or her entire adult life. This questionnaire analyzes the Education, Working Activity and Leisure Time with point subscales based on the years for each activity. The cognitive reserve outcome is valuated as below: low≤ 70, medium-low 70 : 84, medium 85 : 114, medium-high 115 : 130 , high ≥ 130
variations of physical performance (BIA) | Day 0-180-360
  Bioelectrical impedance analysis (BIA)
variations of physical performance (hand grip) | Day 0-180-360
  Hand grip test
variations of physical performance ( timed up and go) | Day 0-180-360
  timed up and go test
variations of physical performance (SPPB) | Day 0-180-360
  Short Physical Performance Battery (SPPB)
variations of physical performance (Frailty index) | Day 0-180-360
  Frailty index was developed to assess for frailty risk in older adults using items collected in existing nursing datasets. This is a questionnaire composed by 10 items and represents an assessment instrument with scores ranging from 0-10. A score of 0 indicates no frailty; a score of 1-3 indicates frailty risk; and a score of 4 or greater indicates frailty
variations of physical performance (ADL) | Day 0-180-360
  Activities of daily living (ADL)
variations of physical performance (IADL) | Day 0-180-360
  Instrumental Activities of Daily Living (IADL)
variations of modification of biochemical parameters of inflammation. | Day 0-180-360
  Measuring circulating levels of inflammation cytokines: EGF, Eotaxin, G-CSF, GM-CSF, IFNα2, IFNγ, IL-10, IL-12P40, IL-12P70, IL-13, IL-15, IL-17A, IL-1RA, IL-1α, IL-1β, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IP-10, MCP-1, MIP-1α, MIP-1β, RANTES, TNFα, TNFβ, VEGF, FGF-2, TGF-α, FIT-3L, Fractalkine, GRO, MCP-3, MDC, PDGF-AA, PDGF-BB, sCD40L, and IL-9.
variations of modification of oxidative stress conditions parameters. | Day 0-180-360
  Measuring circulating levels of E Vitamins, Superoxide dismutase (SOD), catalase, GPx.
variations of changes in the microbiota (bacteria subpopulations) | Day 0-180-360
  to evaluate the potential variations of changes in bacteria populations in the microbiota after 6 and after 12 months of treatment compared to baseline and compared to placebo.
variations of changes in the microbiota (SCFA) | Day 0-180-360
  to evaluate the potential variations of changes in short chain fatty acids levels in the microbiota after 6 and after 12 months of treatment compared to baseline and compared to placebo.
Safety and Tolerability (Adverse Events) | Day 0 to Day 360
  Number of Adverse events and serious adverse events that will be recorded throughout the duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- S.C. di Geriatria Ospedale S. Maria della Misericordia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No